CLINICAL TRIAL: NCT06326879
Title: Early-Onset Colorectal Cancer Versus Late-Onset Colorectal Cancer: a Prospective Observational Cohort Study to Explore the Clinical, Sociodemographic, Genetic, and Molecular Characteristics Associated With Adverse Oncological Outcomes (
Brief Title: A Comparative Study Between Early Onset Colorectal Cancer and Late Onset Colorectal Cancer Patients
Acronym: EOrOS
Status: Recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 3527
Record Dates: First submitted 2024-03-18; First posted 2024-03-22 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer
Keywords: Early Onset Colorectal Cancer; Cancer survival; Genetic and molecular characterization
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples collected before the surgical intervention, and six, twelve, and twenty-four months after surgery; fresh tumor sample collected at surgery; Formalin-Fixed Paraffin-Embedded (FFPE) tumor collected at surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early Onset Colorectal Cancer (EOCRC): Patients aged less or equal to 49 years old at the time of colorectal cancer diagnosis
  Interventions: Other: No intervention
- Late Onset Colorectal Cancer (LOCRC): Patients aged more or equal to 50 years old at the time of colorectal cancer diagnosis
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Questionnaires compilation and sample collection

SUMMARY:
This study aims to investigate the clinical, socioeconomic, behavioral, genetic, and molecular factors characterizing Early Onset Colorectal Cancer (EOCRC) patients compared with Late Onset Colorectal Cancer (LOCRC) patients

DETAILED DESCRIPTION:
Early Onset Colorectal Cancer (EOCRC), defined as a Colorectal Cancer (CRC) arising before the age of 50, is increasing and displays more aggressive features compared with Late Onset Colorectal Cancer (LOCRC, with a diagnosis after the age of 50). EOCRC patients have indeed a higher incidence rate of CRC recurrence after surgery compared with LOCRC, even at early CRC stages (stage I or II). The reasons underlying the more aggressive patterns are almost unknown but may span and can be represented by a combination of socioeconomic factors (including low economic income and access to screening programs, diagnosis, or therapy), behavioral and lifestyle factors (including diet, sedentary behaviors, or increased stress and anxiety), and molecular or genetic factors.

The aim of this study is to prospectively validate our previous retrospective findings, demonstrating a higher incidence rate of CRC recurrence in early stage EOCRC, and explore the possible association between lifestyle, dietary, socioeconomics, molecular and genetic factors and postoperative CRC survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years old at the time of inclusion.
* Patients with a proven diagnosis of colorectal adenocarcinoma, as reported by the staging histological biopsies.
* Patients with a preoperative staging I-III.
* Patients scheduled for elective curative colorectal resection.
* Patients with rectal cancer who underwent neoadjuvant therapy can be included in the study.
* Patients able and willing to comply with the protocol requirements (samples' collection and questionnaires' compilation).

Exclusion Criteria:

* Patients with metastatic disease at diagnosis.
* Patients requiring an emergent procedure.
* Patients undergoing palliative surgery (for example, fecal diversion).
* Patients with a surgical indication for benign lesions (for example, adenoma or dysplasia).
* Patients with an intraoperative finding of a lesion other than adenocarcinoma will be withdrawn from the study.
* Patients with an intraoperative finding of distal metastasis or peritoneal carcinosis will be withdrawn from the study.
* Patients with a concomitant diagnosis of Inflammatory Bowel Disease.
* Patients with a known genetic syndrome (for example, Lynch syndrome or Familial Adenomatous Polyposis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients with a proven diagnosis of stage I-III colorectal adenocarcinoma, scheduled for elective curative cancer resection.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate ratio of colorectal cancer recurrence | 24 months after surgery
  Incidence rate ratio of 24-month colorectal cancer recurrence- defined as any radiological or endoscopic evidence of local recurrence or distal metastasis after the index surgery in stage I-III patients- between the study cohorts

SECONDARY OUTCOMES:
Correlation between lifestyle and incidence rate of colorectal cancer recurrence | 24 months after surgery
  Compare the association between physical activity, dietary, and lifestyle behaviors and 24-month colorectal cancer recurrence in the study cohorts.
Correlation between genetic profile and incidence rate of colorectal cancer recurrence | 24 months after surgery
  Compare the association between the genetic profile of the surgical specimens, as identified by whole exome sequencing of the fresh and paraffin-embedded tumor specimen, and the 24-month CRC recurrence in the study cohorts
Correlation between molecular profile and incidence rate of colorectal cancer recurrence | 24 months after surgery
  Compare the association between the molecular profile of the serum samples and surgical specimens, as identified by RNA sequencing and spatial transcriptomic analyses at different time points during the follow-up, and 24-month CRC recurrence between the study cohorts
Correlation between socioeconomic characteristics and incidence rate of colorectal cancer recurrence | 24 months after surgery
  Compare the association between socioeconomic characteristics, including access to health resources and inclusion in screening programs or experimental therapies, and 24-month CRC recurrence in the study cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Spinelli, MD, PhD, Principal Investigator — IRCCS Huamanitas Research Hospital
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No